CLINICAL TRIAL: NCT01015391
Title: A Randomized, Controlled, Open-label Study to Assess the Efficacy of T2 Versus Azathioprine for the Maintenance of Clinical and Endoscopic Remission in Subjects With Crohn's Disease After Surgical Resection
Brief Title: Efficacy Study of T2 Versus AZA to Maintain Clinical and Endoscopic Remission in Postoperative Crohn's Disease
Acronym: T2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, vice director of General surgery institute, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TW2-001
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Crohn's Disease
Keywords: T2; AZA; remission; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T2 (Experimental)
  Interventions: Drug: T2
- AZA (Active Comparator)
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: T2 — 1.5mg/kg/day, PO (per oral),three times a day: until progression or unacceptable toxicity develops
  Arms: T2
Drug: Azathioprine — 2.5mg/kg, PO (per oral) one time a day:until progression or unacceptable toxicity develops the first month:1.5mg/kg,PO,one time a day the second month:2.0mg/kg,PO,one time a day since the third month:2.5mg/kg,PO,one time a day
  Arms: AZA

SUMMARY:
The purpose of this study is to see whether T2 versus Azathioprine is able to maintain the clinical and endoscopic remission in subjects with Crohn's disease after surgery-induced remission.

The side effects related to T2 and AZA will also be monitored throughout the study.

DETAILED DESCRIPTION:
Crohn's disease is characterized by inflammation and ulceration of the small intestine and colon. Patients commonly experience abdominal pain, diarrhea，malnutrition and malaise which result in decreased quality of life and an increased risk of chronic disability and unemployment. Surgical resection is required in approximately 70% of the patients at some time. However, recurrence of the disease after operation occurs in the majority of patients and is a serious limitation of surgical management. Patients' quality of life is often severely diminished. Currently available therapeutic options for the maintenance of remission in Crohn's disease are inadequate. A clear need exists for well-tolerated drugs that can reliably reduce the risk of a disease relapse.

AZA is classical immunomodulator,often applied to hematologic diseases and immune-related diseases,also the most commonly used drug in the maintenance of remission in Crohn's disease, it is indicated in steroid resistant or dependent patients, in those whose frequency of relapse is >1 per year, in patients after induction of remission with IFX, and in patients whose remission were induced by surgical resection. However, AZA may cause some adverse effects,the most serious adverse effect is leucopenia, which can develop suddenly and unpredictably, though it is rare (around 3%).

T2 is a chloroform/methanol extract Tripterygium wilfordii Hook F (TWHF), the traditional Chinese medicine,used in rheumatoid arthritis and nephritis. It has both immunomodulatory and anti-inflammatory activities.Our previous animal studies have revealed that the major component of T2, triptolide, could prevent the development of chronic colitis in interleukin-10 deficient mice. The phase I clinical trial in our institute also demonstrated that T2, or combined with enteral nutrition, is efficient for induction of remission in patients with active Crohn's disease.The common adverse effects of T2 are leucopenia,liver renal toxicity,oligospermia and amenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have a definitive diagnosis of Crohn's disease, based on WHO criteria
* Subjects having curative resection/ileocolonic anastomosis，pathologically diagnosed as Crohn's disease
* Lesions located in ileum or ileocecal region
* Males and females ≥ 18 years old, including women who are not pregnant or lactating at the time of enrollment.
* Body weight between 40 and 100 kg, inclusive.
* Subjects should have a CDAI score <150 at week 0
* Able to swallow tablets
* Are capable of providing written informed consent and obtained at the time of enrollment
* Willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Bacterial,viral or other microbial infection(including HIV)
* any of the following medications taken within 12 weeks before surgery: cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, or other investigational drugs
* any of ongoing therapy for Crohn's disease with: 5-ASA compounds, steroids, immune modifiers, systemic antibiotics, and tube feeding
* Needing orally administered corticosteroids for the treatment of other diseases. Inhaled or dermatologic preparations are acceptable.
* Previous or current use of infliximab.
* current use of prescription doses or chronic/frequent use of NSAIDs
* Treatment with narcotic pain medications. (Anti-diarrheal agents such as loperamide and diphenoxylate are permitted, providing that the dose is not increased during the study period.)
* With an ileal or colonic stoma.
* History of pancreatitis, except for subjects with a known but removed cause(such as gallstone pancreatitis)
* WBC <3.0 x 109/L, hemoglobin <80 g/L, Platelets<50,000/mm3 at the time of enrollment (or within the previous 6 months, if known)
* History of abnormal liver function tests, including AST or ALT >1.5 times upper limit of normal, alkaline phosphatase >2 times upper limit of normal, total bilirubin >2.5 mg/dL at screening (or within the previous 6 months, if known)
* With short bowel syndrome (defined as requiring oral or parenteral supplemental or total nutrition to maintain stable body weight, or more than 100 cm of small bowel resected)
* History of malignancy
* Women who are pregnant or lactating at the time of enrollment, or who intend to be during the study period.
* Participation in other clinical trial within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission: the proportion of patients with CDAI <150 at 26 and 52 weeks | 52 weeks
Endoscopic Remission: the proportion of patients with CDEIS <6 at 26 and 52 weeks | 52 weeks

SECONDARY OUTCOMES:
The time till the clinical relapse of CD(the CDAI >150 or an increase of more than 70 points) | 52 weeks
The time till the histological recurrence(determined by biopsies and endoscopic findings) | 52 weeks
Serum C-reactive protein concentration; Erythrocyte Sedimentation Rate | 52 weeks
The proportion of patients experiencing adverse events | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Zhu, PhD,MD, Principal Investigator — General Surgery Institute,Jinling Hospital,Nanjing,Jiangsu,China
Locations (1):
- General Surgery Institute,Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Hanauer SB, Korelitz BI, Rutgeerts P, Peppercorn MA, Thisted RA, Cohen RD, Present DH. Postoperative maintenance of Crohn's disease remission with 6-mercaptopurine, mesalamine, or placebo: a 2-year trial. Gastroenterology. 2004 Sep;127(3):723-9. doi: 10.1053/j.gastro.2004.06.002. PMID 15362027
- [Background] Almer SH, Hjortswang H, Hindorf U. 6-Thioguanine therapy in Crohn's disease--observational data in Swedish patients. Dig Liver Dis. 2009 Mar;41(3):194-200. doi: 10.1016/j.dld.2008.07.314. Epub 2008 Sep 16. PMID 18799369
- [Background] Goldbach-Mansky R, Wilson M, Fleischmann R, Olsen N, Silverfield J, Kempf P, Kivitz A, Sherrer Y, Pucino F, Csako G, Costello R, Pham TH, Snyder C, van der Heijde D, Tao X, Wesley R, Lipsky PE. Comparison of Tripterygium wilfordii Hook F versus sulfasalazine in the treatment of rheumatoid arthritis: a randomized trial. Ann Intern Med. 2009 Aug 18;151(4):229-40, W49-51. doi: 10.7326/0003-4819-151-4-200908180-00005. PMID 19687490
- [Background] Peyrin-Biroulet L, Deltenre P, Ardizzone S, D'Haens G, Hanauer SB, Herfarth H, Lemann M, Colombel JF. Azathioprine and 6-mercaptopurine for the prevention of postoperative recurrence in Crohn's disease: a meta-analysis. Am J Gastroenterol. 2009 Aug;104(8):2089-96. doi: 10.1038/ajg.2009.301. Epub 2009 Jun 30. PMID 19568226
- [Background] Ren J, Tao Q, Wang X, Wang Z, Li J. Efficacy of T2 in active Crohn's disease: a prospective study report. Dig Dis Sci. 2007 Aug;52(8):1790-7. doi: 10.1007/s10620-007-9747-y. Epub 2007 Apr 5. PMID 17410440
- [Background] Wei X, Gong J, Zhu J, Niu L, Zhu W, Li N, Li J. Therapeutic effects of triptolide on interleukin-10 gene-deficient mice with colitis. Int Immunopharmacol. 2008 Dec 20;8(13-14):1808-12. doi: 10.1016/j.intimp.2008.08.019. Epub 2008 Sep 17. PMID 18804190
- [Background] Wei X, Gong J, Zhu J, Wang P, Li N, Zhu W, Li J. The suppressive effect of triptolide on chronic colitis and TNF-alpha/TNFR2 signal pathway in interleukin-10 deficient mice. Clin Immunol. 2008 Nov;129(2):211-8. doi: 10.1016/j.clim.2008.07.018. Epub 2008 Aug 30. PMID 18757245
- [Background] Caprilli R, Gassull MA, Escher JC, Moser G, Munkholm P, Forbes A, Hommes DW, Lochs H, Angelucci E, Cocco A, Vucelic B, Hildebrand H, Kolacek S, Riis L, Lukas M, de Franchis R, Hamilton M, Jantschek G, Michetti P, O'Morain C, Anwar MM, Freitas JL, Mouzas IA, Baert F, Mitchell R, Hawkey CJ; European Crohn's and Colitis Organisation. European evidence based consensus on the diagnosis and management of Crohn's disease: special situations. Gut. 2006 Mar;55 Suppl 1(Suppl 1):i36-58. doi: 10.1136/gut.2005.081950c. PMID 16481630
- [Background] Travis SP, Stange EF, Lemann M, Oresland T, Chowers Y, Forbes A, D'Haens G, Kitis G, Cortot A, Prantera C, Marteau P, Colombel JF, Gionchetti P, Bouhnik Y, Tiret E, Kroesen J, Starlinger M, Mortensen NJ; European Crohn's and Colitis Organisation. European evidence based consensus on the diagnosis and management of Crohn's disease: current management. Gut. 2006 Mar;55 Suppl 1(Suppl 1):i16-35. doi: 10.1136/gut.2005.081950b. PMID 16481629
- [Background] Stange EF, Travis SP, Vermeire S, Beglinger C, Kupcinkas L, Geboes K, Barakauskiene A, Villanacci V, Von Herbay A, Warren BF, Gasche C, Tilg H, Schreiber SW, Scholmerich J, Reinisch W; European Crohn's and Colitis Organisation. European evidence based consensus on the diagnosis and management of Crohn's disease: definitions and diagnosis. Gut. 2006 Mar;55 Suppl 1(Suppl 1):i1-15. doi: 10.1136/gut.2005.081950a. No abstract available. PMID 16481628